CLINICAL TRIAL: NCT00318032
Title: A Randomised Trial of the Cost Effectiveness of Screening and Intensive Multi-factorial Intervention for Type 2 Diabetes
Brief Title: A Study to Investigate the Benefits of the Early Detection and Intensive Treatment of Type 2 Diabetes
Acronym: ADDITION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Department of Health, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 9320; 7254
Record Dates: First submitted 2006-01-23; First posted 2006-04-25 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Randomised control trial; Screening; Intensive management; Diabetes mellitus; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

ARMS (1):
- Intensive Treatment (Other): Frequent specialised diabetes clinician contact. DESMOND self-management programme
  Interventions: Drug: multi-factorial intervention

INTERVENTIONS:
Drug: multi-factorial intervention

SUMMARY:
Diabetes is a common chronic condition associated with the risk of heart disease, and eye and kidney damage. Many people are diagnosed with diabetes when they develop symptoms or complications, suggesting that the true onset of disease occurs years earlier. Early detection of diabetes may result in health benefits, but this is not proven. People of South Asian origin are at more risk of having diabetes and of getting the heart disease complications associated with it. The study aims to test whether screening for diabetes is feasible in a South Asian population and to measure the benefits of early detection and intensive treatment.

Hypothesis: A program of screening and an intensive multi-factorial intervention for type 2 diabetes is both feasible and cost effective within primary care.

DETAILED DESCRIPTION:
Although diabetes is commonly undiagnosed and many patients have evidence of complications at diagnosis, there is no definitive evidence that early detection improves health outcomes. One of the critical but uncertain factors is the extent to which screening and subsequent treatment reduces cardiovascular risk. Multi-factorial cardiovascular risk reduction in people with prevalent diabetes and microalbuminuria results in a halving of heart disease risk. However, it is not certain whether this result can be generalised to patients without microalbuminuria or those whose disease is screen-detected.

The ADDITION study is a collaborative randomised controlled trial of a target-driven intensive multi-factorial approach to cardiovascular risk reduction in patients with screen-detected type 2 diabetes mellitus, aimed at assessing the feasibility of screening in a primary care setting and quantifying the cardiovascular benefits and economic and psychological costs of screening. The study as a whole will have the power to determine whether screening and the intensive multi-factorial intervention results in improved cardiovascular outcomes. The ADDITON-Leicester study will contribute to this collaboration, but which by itself will demonstrate the feasibility of screening and measure the effect of the ADDITION study intervention on modelled cardiovascular risk at 1 year after detection by screening in a population at high risk by virtue of having a high proportion of people from South Asia (Leicester). The study is also assessing the impact of intensive intervention of modelled cardiovascular risk at 1 year.

People of South Asian origin are at increased risk of having diabetes and of developing heart disease. The issues of screening are thus particularly relevant to this population. However, all of the populations currently recruited to ADDITION are predominantly Caucasian. The ADDITION-Leicester study will assess the feasibility of systematic screening in a South Asian population, will quantify the effect of intensive treatment in people with screen detected diabetes on modelled cardiovascular risk at 1 year and will assess the economic and psychological costs of screening and intensive treatment. This study population will then contribute to the ADDITION-Europe study, which as a whole is powered to assess the impact of screening and intensive treatment on 5 year cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients who will be included into the study will be from the following groups:

* White European subjects aged between 40-75 years
* Asian, Black, or Chinese subjects aged between 25-75 years

Exclusion Criteria:

Patients will be excluded from the study if they:

* Are housebound
* Have a terminal illness
* Have diabetes mellitus
* Have an active psychotic illness which deems them unable to give informed consent.
* Are pregnant or lactating
* Are taking part in any other clinical trials

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8579 (Actual)
Dates: Start 2004-08; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
To contribute to the ADDITION-Europe study, to assess screening and intensive treatment on 5 year cardiovascular outcomes | At end of study

SECONDARY OUTCOMES:
To assess the feasibility of screening in a South Asian population and the effect of intensive treatment in people with screen detected diabetes on modelled cardiovascular risk at 1 year | At end of study
To assess the economic and psychological cost of screening | At end of study

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester Royal Infirmary, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Peer N, Balakrishna Y, Durao S. Screening for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 May 29;5(5):CD005266. doi: 10.1002/14651858.CD005266.pub2. PMID 32470201
- [Derived] Webb D, Dales J, Zaccardi F, Hill S, Moore C, Farooqi A, Griffin S, Davies M, Khunti K. Intensive versus standard multifactorial cardiovascular risk factor control in screen-detected type 2 diabetes: 5-year and longer-term modelled outcomes of the ADDITION-Leicester study. Diabetes Metab Res Rev. 2019 Mar;35(3):e3111. doi: 10.1002/dmrr.3111. Epub 2018 Dec 19. PMID 30521699
- [Derived] Kidy FF, Dhalwani N, Harrington DM, Gray LJ, Bodicoat DH, Webb D, Davies MJ, Khunti K. Associations Between Anthropometric Measurements and Cardiometabolic Risk Factors in White European and South Asian Adults in the United Kingdom. Mayo Clin Proc. 2017 Jun;92(6):925-933. doi: 10.1016/j.mayocp.2017.02.009. PMID 28578782
- [Derived] Bodicoat DH, O'Donovan G, Dalton AM, Gray LJ, Yates T, Edwardson C, Hill S, Webb DR, Khunti K, Davies MJ, Jones AP. The association between neighbourhood greenspace and type 2 diabetes in a large cross-sectional study. BMJ Open. 2014 Dec 23;4(12):e006076. doi: 10.1136/bmjopen-2014-006076. PMID 25537783
- [Derived] Mostafa SA, Davies MJ, Morris DH, Yates T, Srinivasan BT, Webb D, Brady E, Khunti K. The association of the triglyceride-to-HDL cholesterol ratio with insulin resistance in White European and South Asian men and women. PLoS One. 2012;7(12):e50931. doi: 10.1371/journal.pone.0050931. Epub 2012 Dec 10. PMID 23251403
- [Derived] Mostafa SA, Khunti K, Kilpatrick ES, Webb D, Srinivasan BT, Gray LJ, Davies MJ. Diagnostic performance of using one- or two-HbA1c cut-point strategies to detect undiagnosed type 2 diabetes and impaired glucose regulation within a multi-ethnic population. Diab Vasc Dis Res. 2013 Jan;10(1):84-92. doi: 10.1177/1479164112451473. Epub 2012 Jul 6. PMID 22773521
- [Derived] Mostafa SA, Davies MJ, Webb DR, Srinivasan BT, Gray LJ, Khunti K. Independent effect of ethnicity on glycemia in South Asians and white Europeans. Diabetes Care. 2012 Aug;35(8):1746-8. doi: 10.2337/dc11-2079. Epub 2012 Jun 14. PMID 22699291
- [Derived] Gray LJ, Yates T, Davies MJ, Brady E, Webb DR, Sattar N, Khunti K. Defining obesity cut-off points for migrant South Asians. PLoS One. 2011;6(10):e26464. doi: 10.1371/journal.pone.0026464. Epub 2011 Oct 19. PMID 22039493
- [Derived] Webb DR, Gray LJ, Khunti K, Srinivasan B, Taub N, Campbell S, Barnett J, Farooqi A, Echouffo-Tcheugui JB, Griffin SJ, Wareham NJ, Davies MJ. Screening for diabetes using an oral glucose tolerance test within a western multi-ethnic population identifies modifiable cardiovascular risk: the ADDITION-Leicester study. Diabetologia. 2011 Sep;54(9):2237-46. doi: 10.1007/s00125-011-2189-2. Epub 2011 Jun 3. PMID 21638133
- [Derived] Webb DR, Khunti K, Srinivasan B, Gray LJ, Taub N, Campbell S, Barnett J, Henson J, Hiles S, Farooqi A, Griffin SJ, Wareham NJ, Davies MJ. Rationale and design of the ADDITION-Leicester study, a systematic screening programme and randomised controlled trial of multi-factorial cardiovascular risk intervention in people with type 2 diabetes mellitus detected by screening. Trials. 2010 Feb 19;11:16. doi: 10.1186/1745-6215-11-16. PMID 20170482